CLINICAL TRIAL: NCT04712058
Title: A Multicenter Clinical Trial to Evaluate the Feasibility and Outcome of Same-day Antiretroviral Therapy With Bictegravir/Emtricitabine/Tenofovir Alafenamide (BIC/F/TAF) Among Patients Testing Positive by HIV Confirmatory Tests
Brief Title: Same-day Antiretroviral Therapy With BIC/F/TAF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Far Eastern Memorial Hospital (Other); Mackay Memorial Hospital (Other); Changhua Christian Hospital (Other); Chung Shan Medical University (Other); National Cheng-Kung University Hospital (Other); Chi Mei Medical Hospital (Other); Kaohsiung Medical University Chung-Ho Memorial Hospital (Other); Kaohsiung Municipal Ta-Tung Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202003020MIPB
Record Dates: First submitted 2021-01-14; First posted 2021-01-15 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2020-12

CONDITIONS: HIV Infections
Keywords: same-day initiation, rapid initiation
MeSH Terms: conditions — HIV Infections | interventions — bictegravir; Emtricitabine; tenofovir alafenamide; bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Same-day initiation with BIC/F/TAF (Experimental)
  Interventions: Drug: Bictegravir / Emtricitabine / Tenofovir Alafenamide Oral Tablet [Biktarvy]

INTERVENTIONS:
Drug: Bictegravir / Emtricitabine / Tenofovir Alafenamide Oral Tablet [Biktarvy] — Biktarvy will be administered on the same day of diagnosis. The daily dosing will be continued for 48 weeks.

SUMMARY:
WHO had recommened rapid ART initiation, defined as starting ART within 7 days or on the same day after HIV diagnosis, to improve HIV care continuum. Prior studies revealed that point-of-care diagnostic methods for the detection of HIV RNA can accelerate linkage to care and reduce anxiety. By shortening the interval between infectious disease physician referral, time-lag between screening and confirmatory tests, with the use of the newly developed point-of-care immunochromatographic confirmatory test, initiating a safe and potent antiretroviral therapy, BIC/F/TAF, on the same day of HIV confirmation will be feasible to improve linkage to care and to shorten the interval between HIV diagnosis and viral suppression.

DETAILED DESCRIPTION:
Background In 2015, WHO recommended that all patients be treated with combination antiretroviral therapy (cART) once the diagnosis of HIV infection was made. On the population level, starting cART soon after HIV diagnosis can prevent onward HIV transmission. Although WHO has recommended "treat-all" policy since 2015, there were still 1.8 million people becoming newly infected with HIV in 20179. The substantial loss of patients during the HIV care continuum among the most vulnerable populations have been major concerns in the cART scale-up. Therefore, the concept of rapid ART initiation, defined as starting ART within 7 days or even on the same day after HIV diagnosis was confirmed, was introduced to improve HIV care continuum. In several clinical trials, loss to follow-up was observed despite the clinical trial settings. From our prior study18, among 786 individuals who were screened positive for HIV, 2.4% never returned to the clinic for the confirmatory tests. Despite ART scale-up and the policy of rapid initiation, 30% the of patients who were diagnosed with HIV infection during 2017-2018 did not initiate cART within 7 days after HIV diagnosis was made. Prior studies revealed that point-of-care diagnostic methods for detection of HIV RNA can accelerate linkage to care and reduce anxiety. However, the cost of and the barriers to accessing the point-of-care HIV RNA testing remain high. By shortening the interval between infectious disease physician referral, time-lag between screening and confirmatory tests, with the use of newly developed point-of-care immunochromatographic confirmatory test, initiating a safe and potent antiretroviral therapy on the same day of HIV confirmation will be feasible to improve linkage to care and to shorten the interval between HIV diagnosis and viral suppression.

Study aim This study objective is to investigate the feasibility and outcomes of same-day initiation with Biktarvy (Bic/F/TAF) among patients who receive a diagnosis of HIV infection by confirmatory test.

Study Interventions This is a multi-center, single-arm, prospective cohort study. All individuals who fulfill the inclusion/exclusion criteria will be enrolled in our study and followed for 48 weeks. During the first visit at ID clinic, baseline clinical data will be collected by history taking, physical examination, and blood testing. The confirmatory test and baseline evaluations will be performed at the Visit 1. The test results will also be reported on the same day. Patients, who are HIV(+) by confirmatory test ,will receive a 7-day Biktarvy treatment and the first dose will be administered from Visit 1 (Day 1). The results of other evaluation including viral load, CD4 count, and coinfection will be available at visit 2.

At Visit 2, the clinical symptoms and the tolerability will be recorded. If participants continue to receive Biktarvy® at the discretion of the HIV treating physicians, Biktarvy will be continued according to the national HIV treatment guidelines, which will be reimbursed by the National Health Insurance, and the patients will be followed in our study for 48 weeks. If the patients are switched to other cART regimens than Bictarvy according to physician's clinical judgements, the participants will continue their follow-up in the study.

During the follow-up period, clinical information on symptoms, tolerability, and adverse effects with the use of face-to-face questionnaire interviews, and follow-up laboratory test results will be collected. to evaluate the efficacy and adverse effect according to the national HIV treatment guidelines and routine clinical practices.

Monitor of Adverse event and management The subjective adverse events will be inquired during each visit and recorded with the use of questionnaire interviews. According to the national HIV treatment guidelines in Taiwan, the liver and renal functions and muscle enzymes will be followed during treatment as part of the standard of care. The study team will provide best clinical care if adverse events develop and the cost of medical care required will be covered by the insurance company. Severe adverse event and withdrawal from the study will be reported to the primary investigator on a monthly basis. When the number of drop-out is higher than 30%, the enrollment will be stopped temporarily until the investigation ensures the safety of the participants.

Study Endpoints

1. Primary endpoints 1) The rate of retention in care at Week 48 2) The proportion of viral suppression (<50 copies/ml) at Week 48
2. Secondary endpoints 1) The rate of same-day initiation of ART among patients who receive a confirmed diagnosis of HIV infection 2) The proportion of viral suppression (<200 copies/ml) at Weeks 1, 4, and 48 3) Any/severe adverse effect of B/F/TAF before Weeks 4 and 48 4) Patient's satisfaction at Weeks 1, 4, and 48

Statistical analysis

1. This is a feasibility study aiming to investigate the rate of engagement in same-day ART initiation and retention in care at Week 48. No sample size calculation is needed. The sample size of 200 participants is estimated by taking into account the case numbers of newly diagnosed HIV-positive patients seeking HIV care and cART at each participating hospitals during the past 1 year.
2. Timetable for study and enrollment:

1) Total subjects expected to be enrolled: 200 2) Total subjects expected to enter treatment: 195 3) Total subjects expected to complete treatment: 191 4) Duration of enrolled period: 20 months 5) Number of subjects entering treatment per month: 10 ( 2 subjects per site)

ELIGIBILITY:
Inclusion Criteria:

* Patients who test positive by HIV screening tests (4th generation Ag/Ab) by clinical care providers or by VCT counselors within 3 days of Visit 1.
* Aged 20 years or older
* Patient is willing to participate in this study and sign the written informed consent form

Exclusion Criteria:

* Prior HIV diagnosis
* Prior ART for HIV infection
* Chronic kidney disease, stage ≥4 (CCr <30 ml/min/1.73m2) or receiving dialysis
* Severe hepatic impairment (Child-Pugh score C) or clinical apparent hepatic impairment including jaundice or ascites
* Active or latent tuberculosis infection or clinical apparent central nervous system infection
* Pregnancy or breastfeeding
* Allergy to FTC or TDF containing medication

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-01-20 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Retention in care at Week 48 | week 48 ± 4wk
  The proportion of patients who returned for the scheduled clinic visit at week 48
Viral suppression at Week 48 | week 48 ± 4wk
  The proportion of viral suppression (<50 copies/ml) at week 48

SECONDARY OUTCOMES:
Acceptability of same-day initiation | Day 1
  The rate of same-day initiation of ART among patients who receive a confirmed diagnosis of HIV infection
Viral suppression at Week 1, 4, 48 | Week 1 ± 3 days, Week 4± 1 week, Week 48± 4 week
  The proportion of viral suppression (<200 copies/ml) at Week 1, 4, 48
Adverse effect at Week 4 and 48 | Week 4± 1 week, Week 48± 4 week
  Any/severe adverse effect of B/F/TAF before Weeks 4 and 48
Patient's satisfaction at Weeks 1, 4, and 48 | Week 1 ± 3 days, Week 4± 1 week, Week 48± 4 week
  Patient's satisfaction with HIV Treatment Satisfaction Questionnaire at Weeks 1, 4, and 48

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] TEMPRANO ANRS 12136 Study Group; Danel C, Moh R, Gabillard D, Badje A, Le Carrou J, Ouassa T, Ouattara E, Anzian A, Ntakpe JB, Minga A, Kouame GM, Bouhoussou F, Emieme A, Kouame A, Inwoley A, Toni TD, Ahiboh H, Kabran M, Rabe C, Sidibe B, Nzunetu G, Konan R, Gnokoro J, Gouesse P, Messou E, Dohoun L, Kamagate S, Yao A, Amon S, Kouame AB, Koua A, Kouame E, Ndri Y, Ba-Gomis O, Daligou M, Ackoundze S, Hawerlander D, Ani A, Dembele F, Kone F, Guehi C, Kanga C, Koule S, Seri J, Oyebi M, Mbakop N, Makaila O, Babatunde C, Babatounde N, Bleoue G, Tchoutedjem M, Kouadio AC, Sena G, Yededji SY, Assi R, Bakayoko A, Mahassadi A, Attia A, Oussou A, Mobio M, Bamba D, Koman M, Horo A, Deschamps N, Chenal H, Sassan-Morokro M, Konate S, Aka K, Aoussi E, Journot V, Nchot C, Karcher S, Chaix ML, Rouzioux C, Sow PS, Perronne C, Girard PM, Menan H, Bissagnene E, Kadio A, Ettiegne-Traore V, Moh-Semde C, Kouame A, Massumbuko JM, Chene G, Dosso M, Domoua SK, N'Dri-Yoman T, Salamon R, Eholie SP, Anglaret X. A Trial of Early Antiretrovirals and Isoniazid Preventive Therapy in Africa. N Engl J Med. 2015 Aug 27;373(9):808-22. doi: 10.1056/NEJMoa1507198. Epub 2015 Jul 20. PMID 26193126
- [Background] INSIGHT START Study Group; Lundgren JD, Babiker AG, Gordin F, Emery S, Grund B, Sharma S, Avihingsanon A, Cooper DA, Fatkenheuer G, Llibre JM, Molina JM, Munderi P, Schechter M, Wood R, Klingman KL, Collins S, Lane HC, Phillips AN, Neaton JD. Initiation of Antiretroviral Therapy in Early Asymptomatic HIV Infection. N Engl J Med. 2015 Aug 27;373(9):795-807. doi: 10.1056/NEJMoa1506816. Epub 2015 Jul 20. PMID 26192873
- [Background] O'Connor J, Vjecha MJ, Phillips AN, Angus B, Cooper D, Grinsztejn B, Lopardo G, Das S, Wood R, Wilkin A, Klinker H, Kantipong P, Klingman KL, Jilich D, Herieka E, Denning E, Abubakar I, Gordin F, Lundgren JD; INSIGHT START study group. Effect of immediate initiation of antiretroviral therapy on risk of severe bacterial infections in HIV-positive people with CD4 cell counts of more than 500 cells per muL: secondary outcome results from a randomised controlled trial. Lancet HIV. 2017 Mar;4(3):e105-e112. doi: 10.1016/S2352-3018(16)30216-8. Epub 2017 Jan 5. PMID 28063815
- [Background] Guideline on When to Start Antiretroviral Therapy and on Pre-Exposure Prophylaxis for HIV. Geneva: World Health Organization; 2015 Sep. Available from http://www.ncbi.nlm.nih.gov/books/NBK327115/ PMID 26598776
- [Background] Cohen MS, Chen YQ, McCauley M, Gamble T, Hosseinipour MC, Kumarasamy N, Hakim JG, Kumwenda J, Grinsztejn B, Pilotto JH, Godbole SV, Chariyalertsak S, Santos BR, Mayer KH, Hoffman IF, Eshleman SH, Piwowar-Manning E, Cottle L, Zhang XC, Makhema J, Mills LA, Panchia R, Faesen S, Eron J, Gallant J, Havlir D, Swindells S, Elharrar V, Burns D, Taha TE, Nielsen-Saines K, Celentano DD, Essex M, Hudelson SE, Redd AD, Fleming TR; HPTN 052 Study Team. Antiretroviral Therapy for the Prevention of HIV-1 Transmission. N Engl J Med. 2016 Sep 1;375(9):830-9. doi: 10.1056/NEJMoa1600693. Epub 2016 Jul 18. PMID 27424812
- [Background] Rodger AJ, Cambiano V, Bruun T, Vernazza P, Collins S, Degen O, Corbelli GM, Estrada V, Geretti AM, Beloukas A, Raben D, Coll P, Antinori A, Nwokolo N, Rieger A, Prins JM, Blaxhult A, Weber R, Van Eeden A, Brockmeyer NH, Clarke A, Del Romero Guerrero J, Raffi F, Bogner JR, Wandeler G, Gerstoft J, Gutierrez F, Brinkman K, Kitchen M, Ostergaard L, Leon A, Ristola M, Jessen H, Stellbrink HJ, Phillips AN, Lundgren J; PARTNER Study Group. Risk of HIV transmission through condomless sex in serodifferent gay couples with the HIV-positive partner taking suppressive antiretroviral therapy (PARTNER): final results of a multicentre, prospective, observational study. Lancet. 2019 Jun 15;393(10189):2428-2438. doi: 10.1016/S0140-6736(19)30418-0. Epub 2019 May 2. PMID 31056293
- [Background] Minn AC, Kyaw NTT, Aung TK, Mon OM, Htun T, Oo MM, Moe J, Mon AA, Satyanarayana S, Oo HN. Attrition among HIV positive children enrolled under integrated HIV care programme in Myanmar: 12 years cohort analysis. Glob Health Action. 2018;11(1):1510593. doi: 10.1080/16549716.2018.1510593. PMID 30191749
- [Background] Rosen S, Fox MP. Retention in HIV care between testing and treatment in sub-Saharan Africa: a systematic review. PLoS Med. 2011 Jul;8(7):e1001056. doi: 10.1371/journal.pmed.1001056. Epub 2011 Jul 19. PMID 21811403
- [Background] Guidelines for Managing Advanced HIV Disease and Rapid Initiation of Antiretroviral Therapy. Geneva: World Health Organization; 2017. No abstract available. Available from http://www.ncbi.nlm.nih.gov/books/NBK475977/ PMID 29341560
- [Background] Pilcher CD, Ospina-Norvell C, Dasgupta A, Jones D, Hartogensis W, Torres S, Calderon F, Demicco E, Geng E, Gandhi M, Havlir DV, Hatano H. The Effect of Same-Day Observed Initiation of Antiretroviral Therapy on HIV Viral Load and Treatment Outcomes in a US Public Health Setting. J Acquir Immune Defic Syndr. 2017 Jan 1;74(1):44-51. doi: 10.1097/QAI.0000000000001134. PMID 27434707
- [Background] Amanyire G, Semitala FC, Namusobya J, Katuramu R, Kampiire L, Wallenta J, Charlebois E, Camlin C, Kahn J, Chang W, Glidden D, Kamya M, Havlir D, Geng E. Effects of a multicomponent intervention to streamline initiation of antiretroviral therapy in Africa: a stepped-wedge cluster-randomised trial. Lancet HIV. 2016 Nov;3(11):e539-e548. doi: 10.1016/S2352-3018(16)30090-X. Epub 2016 Aug 27. PMID 27658873
- [Background] Rosen S, Maskew M, Fox MP, Nyoni C, Mongwenyana C, Malete G, Sanne I, Bokaba D, Sauls C, Rohr J, Long L. Initiating Antiretroviral Therapy for HIV at a Patient's First Clinic Visit: The RapIT Randomized Controlled Trial. PLoS Med. 2016 May 10;13(5):e1002015. doi: 10.1371/journal.pmed.1002015. eCollection 2016 May. PMID 27163694
- [Background] Malloch L, Kadivar K, Putz J, Levett PN, Tang J, Hatchette TF, Kadkhoda K, Ng D, Ho J, Kim J. Comparative evaluation of the Bio-Rad Geenius HIV-1/2 Confirmatory Assay and the Bio-Rad Multispot HIV-1/2 Rapid Test as an alternative differentiation assay for CLSI M53 algorithm-I. J Clin Virol. 2013 Dec;58 Suppl 1:e85-91. doi: 10.1016/j.jcv.2013.08.008. Epub 2013 Aug 28. PMID 24342484
- [Background] Moon HW, Huh HJ, Oh GY, Lee SG, Lee A, Yun YM, Hur M. Evaluation of the Bio-Rad Geenius HIV 1/2 Confirmation Assay as an Alternative to Western Blot in the Korean Population: A Multi-Center Study. PLoS One. 2015 Sep 30;10(9):e0139169. doi: 10.1371/journal.pone.0139169. eCollection 2015. PMID 26422281
- [Background] Tinguely C, Schild-Spycher T, Bahador Z, Gowland P, Stolz M, Niederhauser C. Comparison of a conventional HIV 1/2 line immunoassay with a rapid confirmatory HIV 1/2 assay. J Virol Methods. 2014 Sep;206:1-4. doi: 10.1016/j.jviromet.2014.05.010. Epub 2014 May 27. PMID 24877900
- [Background] Misumi J, Gardes J, Gonzalez MF, Corvol P, Menard J. Angiotensinogen's role in ANG formation, renin release, and renal hemodynamics in isolated perfused kidney. Am J Physiol. 1989 Apr;256(4 Pt 2):F719-27. doi: 10.1152/ajprenal.1989.256.4.F719. PMID 2539750
- [Background] Gallant J, Lazzarin A, Mills A, Orkin C, Podzamczer D, Tebas P, Girard PM, Brar I, Daar ES, Wohl D, Rockstroh J, Wei X, Custodio J, White K, Martin H, Cheng A, Quirk E. Bictegravir, emtricitabine, and tenofovir alafenamide versus dolutegravir, abacavir, and lamivudine for initial treatment of HIV-1 infection (GS-US-380-1489): a double-blind, multicentre, phase 3, randomised controlled non-inferiority trial. Lancet. 2017 Nov 4;390(10107):2063-2072. doi: 10.1016/S0140-6736(17)32299-7. Epub 2017 Aug 31. PMID 28867497
- [Result] Borges AH, Neuhaus J, Babiker AG, Henry K, Jain MK, Palfreeman A, Mugyenyi P, Domingo P, Hoffmann C, Read TR, Pujari S, Meulbroek M, Johnson M, Wilkin T, Mitsuyasu R; INSIGHT START Study Group. Immediate Antiretroviral Therapy Reduces Risk of Infection-Related Cancer During Early HIV Infection. Clin Infect Dis. 2016 Dec 15;63(12):1668-1676. doi: 10.1093/cid/ciw621. Epub 2016 Sep 8. PMID 27609756
- [Result] Labhardt ND, Ringera I, Lejone TI, Klimkait T, Muhairwe J, Amstutz A, Glass TR. Effect of Offering Same-Day ART vs Usual Health Facility Referral During Home-Based HIV Testing on Linkage to Care and Viral Suppression Among Adults With HIV in Lesotho: The CASCADE Randomized Clinical Trial. JAMA. 2018 Mar 20;319(11):1103-1112. doi: 10.1001/jama.2018.1818. PMID 29509839
- [Result] Langwenya N, Phillips TK, Brittain K, Zerbe A, Abrams EJ, Myer L. Same-day antiretroviral therapy (ART) initiation in pregnancy is not associated with viral suppression or engagement in care: A cohort study. J Int AIDS Soc. 2018 Jun;21(6):e25133. doi: 10.1002/jia2.25133. PMID 29939483
- [Result] Huang YC, Sun HY, Chuang YC, Huang YS, Lin KY, Huang SH, Chen GJ, Luo YZ, Wu PY, Liu WC, Hung CC, Chang SC. Short-term outcomes of rapid initiation of antiretroviral therapy among HIV-positive patients: real-world experience from a single-centre retrospective cohort in Taiwan. BMJ Open. 2019 Sep 20;9(9):e033246. doi: 10.1136/bmjopen-2019-033246. PMID 31542770
- [Result] Wohl D, Clarke A, Maggiolo F, Garner W, Laouri M, Martin H, Quirk E. Patient-Reported Symptoms Over 48 Weeks Among Participants in Randomized, Double-Blind, Phase III Non-inferiority Trials of Adults with HIV on Co-formulated Bictegravir, Emtricitabine, and Tenofovir Alafenamide versus Co-formulated Abacavir, Dolutegravir, and Lamivudine. Patient. 2018 Oct;11(5):561-573. doi: 10.1007/s40271-018-0322-8. PMID 29956087
- [Result] Halperin J, Butler I, Conner K, Myers L, Holm P, Bartram L, Van Sickels N. Linkage and Antiretroviral Therapy Within 72 Hours at a Federally Qualified Health Center in New Orleans. AIDS Patient Care STDS. 2018 Feb;32(2):39-41. doi: 10.1089/apc.2017.0309. No abstract available. PMID 29432044
- [Result] Girometti N, Nwokolo N, McOwan A, Whitlock G. Outcomes of acutely HIV-1-infected individuals following rapid antiretroviral therapy initiation. Antivir Ther. 2017;22(1):77-80. doi: 10.3851/IMP3080. Epub 2016 Sep 2. PMID 27585954
- [Result] Koenig SP, Dorvil N, Devieux JG, Hedt-Gauthier BL, Riviere C, Faustin M, Lavoile K, Perodin C, Apollon A, Duverger L, McNairy ML, Hennessey KA, Souroutzidis A, Cremieux PY, Severe P, Pape JW. Same-day HIV testing with initiation of antiretroviral therapy versus standard care for persons living with HIV: A randomized unblinded trial. PLoS Med. 2017 Jul 25;14(7):e1002357. doi: 10.1371/journal.pmed.1002357. eCollection 2017 Jul. PMID 28742880
- [Result] Stevens WS, Gous NM, MacLeod WB, Long LC, Variava E, Martinson NA, Sanne I, Osih R, Scott LE. Multidisciplinary Point-of-Care Testing in South African Primary Health Care Clinics Accelerates HIV ART Initiation but Does Not Alter Retention in Care. J Acquir Immune Defic Syndr. 2017 Sep 1;76(1):65-73. doi: 10.1097/QAI.0000000000001456. PMID 28542080
- [Result] Meulbroek M, Pujol F, Perez F, Dalmau-Bueno A, Taboada H, Marazzi G, Carrillo A, Cabas A, Gata A, Aldabo E, Roldan B, Coll P, Anez F, Pantaleon J, Mochales M, Gomez V, Marin O, Mir JF, Decoca J, Saz J. BCN Checkpoint: same-day confirmation of reactive HIV rapid test with Point Of Care HIV-RNA accelerates linkage to care and reduces anxiety. HIV Med. 2018 Feb;19 Suppl 1:63-65. doi: 10.1111/hiv.12595. PMID 29488706